CLINICAL TRIAL: NCT00000700
Title: A Multi-Center Clinical Trial To Evaluate Azidothymidine (AZT) in the Treatment of Human Immunodeficiency Virus (HIV) Infection in Patients With AIDS Post First Episode PCP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 002; 10978 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: United States; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To examine the dose of zidovudine (AZT) that was used in the first placebo-controlled study of AZT in AIDS patients as well as a lower dose of AZT in order to determine if the lower dose results in less harmful side effects while still being effective. Previous studies have shown the effectiveness of AZT in AIDS therapy. AZT has been effective in test tube studies at varying doses. There is a need to see if lower doses result in effective therapy with less harmful side effects.

DETAILED DESCRIPTION:
Previous studies have shown the effectiveness of AZT in AIDS therapy. AZT has been effective in test tube studies at varying doses. There is a need to see if lower doses result in effective therapy with less harmful side effects.

Patients are assigned at random to one of two treatment programs: (1) 1 dose of AZT given orally (PO) for 6 doses per day; (2) 2 doses of AZT PO for 4 weeks followed by 1 dose PO for the remainder of the trial.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* All concomitant medication to minimum and record.
* Any approved medications can be used to treat an opportunistic infection.
* Dapsone may be used for Pneumocystis carinii pneumonia (PCP).
* Pyrimethamine - sulfadoxine may be used for toxoplasmosis.
* Ganciclovir for cytomegalovirus may be used for maintenance only.
* Prophylactic therapy for PCP.

Concurrent Treatment:

Allowed:

* Local, limited radiation therapy to isolated Kaposi's sarcoma lesions provided total area is < 5 x 5 cm and a 6-MeV electron beam or 90 kV x-ray = or < 3000 rads total is used.

Patients must have:

* HIV seropositivity as confirmed by any federally licensed ELISA test kit.
* Allowed:
* Malignancy in past which has been in complete remission for 1 year without therapy.

Exclusion Criteria

Co-existing Condition:

Patients with active opportunistic infections will be excluded.

Concurrent Medication:

Excluded:

* Aspirin on a regular basis or beyond 72 hours without contacting investigator.
* Cimetidine.
* Flurazepam.
* Indomethacin.
* Ranitidine.
* Probenecid.

Patients with the following are excluded:

* Status post-Pneumocystis carinii pneumonia with symptomatic visceral Kaposi's sarcoma (KS) or progression of KS within the month prior to study entry.
* Other concurrent neoplasms other than basal cell carcinoma of the skin.
* Requiring blood transfusions > once per month. Last transfusion cannot have been given within 7 days of entry.
* Active substance abuse. Unwilling to sign informed consent or to be followed at medical center where enrolled for duration of study and follow-up if necessary.

Prior Medication:

Excluded within 2 weeks of study entry:

* Treatment for acute Pneumocystis carinii pneumonia (PCP).
* Excluded within 30 days of study entry:
* Other antiretroviral agents, immunomodulating agents, or corticosteroids.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiation therapy or cytotoxic chemotherapy for Kaposi's sarcoma.

Required:

* Patients must be at least 2 weeks post- therapy status for acute Pneumocystis carinii pneumonia (PCP).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 482
Dates: Study Completion 1990-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fischl M, Study Chair
Locations (28):
- United States (28):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Fischl M, Parker CB, Pettinelli C, Wulfsohn M, Rasheed S. The efficacy and safety of a lower dose of zidovudine in the treatment of patients with AIDS-associated PCP. Int Conf AIDS. 1990 Jun 20-23;6(1):138 (abstract no ThB20)
- [Background] De Gruttola V, Wulfsohn M, Fischl MA, Tsiatis A. Modeling the relationship between survival and CD4 lymphocytes in patients with AIDS and AIDS-related complex. J Acquir Immune Defic Syndr (1988). 1993 Apr;6(4):359-65. PMID 8095980
- [Background] McMahon DK, Winkelstein A, Armstrong JA, Pazin GJ, Hawk H, Ho M. Zidovudine therapy is associated with an increased capacity of phytohemagglutinin-stimulated cells to express interleukin-2 receptors. Pittsburgh AIDS Clinical Trial Unit. AIDS. 1991 May;5(5):491-6. doi: 10.1097/00002030-199105000-00003. PMID 1863401
- [Background] Richman DD, Grimes JM, Lagakos SW. Effect of stage of disease and drug dose on zidovudine susceptibilities of isolates of human immunodeficiency virus. J Acquir Immune Defic Syndr (1988). 1990;3(8):743-6. PMID 2114476
- [Background] Wulfsohn M, Fischl M, Tsiatis A. Predictors of survival among patients with AIDS receiving zidovudine. Int Conf AIDS. 1992 Jul 19-24;8(2):C314 (abstract no PoC 4419)
- [Background] Rinaldo C, Huang XL, Piazza P, Armstrong J, Rappocciolo G, Pazin G, McMahon D, Gupta P, Fan Z, Zhang Z, et al. Augmentation of cellular immune function during the early phase of zidovudine treatment of AIDS patients. J Infect Dis. 1991 Oct;164(4):638-45. doi: 10.1093/infdis/164.4.638. PMID 1680135
- [Background] Fischl MA, Parker CB, Pettinelli C, Wulfsohn M, Hirsch MS, Collier AC, Antoniskis D, Ho M, Richman DD, Fuchs E, et al. A randomized controlled trial of a reduced daily dose of zidovudine in patients with the acquired immunodeficiency syndrome. The AIDS Clinical Trials Group. N Engl J Med. 1990 Oct 11;323(15):1009-14. doi: 10.1056/NEJM199010113231501. PMID 1977079
- [Background] Unadkat JD, Collier AC, Crosby SS, Cummings D, Opheim KE, Corey L. Pharmacokinetics of oral zidovudine (azidothymidine) in patients with AIDS when administered with and without a high-fat meal. AIDS. 1990 Mar;4(3):229-32. doi: 10.1097/00002030-199003000-00008. PMID 2350441
- [Background] Coombs RW, Collier AC, Allain JP, Nikora B, Leuther M, Gjerset GF, Corey L. Plasma viremia in human immunodeficiency virus infection. N Engl J Med. 1989 Dec 14;321(24):1626-31. doi: 10.1056/NEJM198912143212402. PMID 2511447